CLINICAL TRIAL: NCT03120416
Title: Effect of Resistance Exercise Training on Endothelial Function and Cardiovascular Risk Factors in Patients With Chronic Kidney Disease
Brief Title: Resistance Exercise Training in Chronic Kidney Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Ana C. Ricardo, MD, MPH, MS, Assistant Professor of Medicine, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2016-0421; K23DK094829 (NIH)
Record Dates: First submitted 2017-04-04; First posted 2017-04-19 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Resistance exercise training program (Experimental): Eight exercises will be used to include large upper and lower body muscle groups. The baseline 1 repetition maximum (RM) will be used to set initial training loads. All exercise sessions will be performed under the supervision of an exercise physiologist. Vital signs and body weight will be recorded before each session. The workload during training will be adjusted to reflect 80% of the most recent 1 RM (approximately 8-12 RM set). In addition, patients' workloads will be progressively increased if the patients can lift the weight more than 12 repetitions. Participants will perform three sets of 8-12 repetitions on each machine per session.
  Interventions: Behavioral: Resistance exercise training
- Control (No Intervention): Participants randomized to the control group will be offered an educational brochure regarding exercise published by the NKF.

INTERVENTIONS:
Behavioral: Resistance exercise training — 12-week resistance exercise training program, 2 times per week, 45 min per session. Eight exercises will be used to include large upper and lower body muscle groups (leg press, leg extension, leg curl, chest press, shoulder extension, biceps curl, abdominal crunch and back extension). The baseline one repetition maximum will be used to set initial training loads.
  Arms: Resistance exercise training program

SUMMARY:
The investigators aim to evaluate the feasibility of a resistance exercise training program among individuals with CKD and its impact on endothelial and vascular function.

DETAILED DESCRIPTION:
Resistance exercise training has been shown to improve cardiovascular health including endothelial function in general populations, but studies in patients with chronic kidney disease (CKD) are limited. The investigators aim to evaluate the feasibility and acceptability of a resistance exercise training program among individuals with CKD and its impact on endothelial and vascular function as measured by brachial artery flow-mediated dilation, pulse-wave velocity and carotid artery stiffness. To accomplish this goal the investigators propose to conduct a 12-week pilot randomized controlled trial of twice a week resistance exercise training among 32 adults with CKD. The results of this study will inform the design and implementation of a larger trial evaluating the impact of resistance exercise training on adverse outcomes in patients with CKD including CKD progression.

ELIGIBILITY:
Inclusion Criteria:

* CKD stage 3 or 4 (eGFR 15-60 ml/min/1.73m2)

Exclusion Criteria:

* Currently institutionalized
* Kidney transplant or dialysis
* NY Heart Association class 3-4 heart failure
* Dementia or cognitive impairment
* Unstable angina or coronary revascularization within the last 3 months
* Uncontrolled arrhythmia
* Severe chronic lung disease
* Orthopedic, neurologic or other condition that would preclude resistance exercise training
* Pregnancy
* Uncontrolled hypertension (systolic > 160 mmHg and diastolic >90 mmHg)

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2017-01-25 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
Endothelial function | 3 months
  Measured by brachial artery flow-mediated dilation (FMD)

SECONDARY OUTCOMES:
Vascular function | 3 months
  Measured by pulse wave velocity
Carotid artery stiffness | 3 months
  Measured by non-invasive ultrasound
Self-reported physical activity | 3 months
  Assessed by the MESA (Multiethnic Study of Atherosclerosis) Typical Week Physical Activity Survey
Objectively measured physical activity | 3 months
  Assessed by a physical activity monitor (ActiGraph GT3X+)
Systolic blood pressure | 3 months
  Measured using standard procedures
Serum LDL-cholesterol | 3 months
  Measured using standard procedures
Serum HDL-cholesterol | 3 months
  Measured using standard procedures
Muscle strength | 3 months
  Assessed by the amount of weight lifted in a single chest press and leg press (1 RM).

CONTACTS AND LOCATIONS:
Overall Officials: Ana C Ricardo, MD, Principal Investigator — Assistant Professor of Medicine
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No